CLINICAL TRIAL: NCT05929950
Title: The Role of Autoimmunity and Obesity in Polycystic Ovary Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ola Ahmed Hamed, Assistant lecturer, Sohag University
Other Study IDs: soh-med-23-06-04MD
Record Dates: First submitted 2023-06-19; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-07

CONDITIONS: Polycystic Ovary Syndrome
Keywords: autoimmunity; obesity; Polycystic ovary syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome; Autoimmune Diseases; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with PCOS
- control group

SUMMARY:
The goal of the study is to detect autoantibodies in the serum of the women with PCOS and evaluate the obesity markers to investigate the the role of autoimmunity and obesity in PCOS

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with PCOS according to the Rotterdam (2003) criteria.

Exclusion Criteria:

* Patients with other causes of hyperandrogenism as congenital adrenal hyperplasia, androgen-secreting tumors, Cushing's syndrome, hyperprolactinemia, virilizing ovarian or adrenal tumors and those taking drugs affecting insulin resistance, such as estrogens, oral contraceptives and corticosteroids during the previous three months before the study.

Ages: 12 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — because the study is about polycystic ovary syndrome
Study Population: women
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
measuring serum anti-ovarian, anti-nuclear, anti-double stranded and anti-thyroid antibodies | 3 months after recruitment
  Theses markers will be measured using ELISA technique

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided